CLINICAL TRIAL: NCT03925025
Title: Effectiveness of Calcium Channel Blockade for Organophosphorus and Carbamate Pesticide Poisoning - an Open, Pragmatic, 3-arm RCT Repurposing Two Widely Available Licensed Medicines
Brief Title: Effectiveness of Calcium Channel Blockade for OP and Carbamate Pesticide Poisoning
Acronym: CCBOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Toxicology Society of Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC19003
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-10

CONDITIONS: Anticholinesterase Insecticide Poisoning; Pesticide Poisoning
MeSH Terms: interventions — Magnesium Sulfate; Nimodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Standard therapy
- Magnesium sulfate (Active Comparator): Standard therapy plus magnesium sulfate
  Interventions: Drug: Magnesium Sulfate
- Nimodipine (Active Comparator): Standard therapy plus nimodipine
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Drug: Magnesium Sulfate — Treatment in addition to standard therapy
  Arms: Magnesium sulfate
Drug: Nimodipine — Treatment in addition to standard therapy
  Arms: Nimodipine

SUMMARY:
This study evaluates whether the addition of intravenous magnesium sulphate or nimodipine to standard therapy (supportive care plus for all patients atropine and, for OP insecticide poisoned patients, pralidoxime) benefits patients after acute anticholinesterase self-poisoning with OP or carbamate insecticides.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years or older with suspected OP or carbamate insecticide self-poisoning admitted to medical wards with the cholinergic toxidrome requiring atropine.
* Diagnosis will be made on the basis of the cholinergic toxidrome clinical features (eg. small/pinpoint pupils, bronchorrhoea, sweating) or on the history of atropine administration with beneficial effect. The insecticide involved will be identified where possible from the history, the bottle brought in by the patient or relative, the patient/relative identifying the pesticide on a chart showing all locally available pesticides, and/or relatives sending a photo of the bottle by eg. WhatsApp.
* Patients who ingest combination products containing OP or carbamate insecticides will also be included.
* Inhibited blood cholinesterase activity as shown by routine clinical bedside test

Exclusion Criteria:

* Children aged <16 years.
* Patients who do not require atropine and have not had it prior to presentation during this episode.
* Normal blood cholinesterase activity
* Self-reported known pregnancy (as per South Asian practice, no attempt will be made to formally test for pregnancy in the patients due to the issue of confidentiality in the acute care situation in these hospitals and the social consequences of an unexpected positive response)
* Known occupational and homicidal poisoning
* Past medical history of severely impaired renal function
* Hypersensitivity to magnesium and its salts
* Patients who have had a myocardial infarction or unstable angina in the last month
* Patients with traumatic subarachnoid haemorrhage
* Lack of informed consent (unaccompanied unconscious patients and others)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1728 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Mortality | through to hospital discharge, median 1 week
  Whether dead or alive at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Dr Fazle Rabbi Chowdhury, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (7):
- Bangladesh (7):
  - Rajshahi Medical College Hospital, Rajshahi, Rajshahi Division
  - Shaheed Ziaur Rahman Medical College, Bogra, Silimpur
  - Chattogram Medical College Hospital, Chittagong
  - Jashore Medical College Hospital, Jessore
  - Khulna Medical College Hospital, Khulna
  - Rangpur Medical College Hospital, Rangpur City
  - Sylhet MAG Osmani Medical College Hospital, Sylhet

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after primary data analysis is published
Access Criteria: From academic group with clear analysis plan

REFERENCES:
- [Background] Brvar M, Chan MY, Dawson AH, Ribchester RR, Eddleston M. Magnesium sulfate and calcium channel blocking drugs as antidotes for acute organophosphorus insecticide poisoning - a systematic review and meta-analysis. Clin Toxicol (Phila). 2018 Aug;56(8):725-736. doi: 10.1080/15563650.2018.1446532. Epub 2018 Mar 20. PMID 29557685